CLINICAL TRIAL: NCT03247920
Title: Intravenous to Oral Antibiotic Switch Therapy for Probable Neonatal Bacterial Infections: Clinical Efficacy, Safety and Cost-effectiveness
Brief Title: Reduction of Intravenous Antibiotics In Neonates
Acronym: RAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Gerdien Tramper, Principal investigator, MD, PhD, Franciscus Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAIN
Record Dates: First submitted 2017-07-03; First posted 2017-08-14 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Neonatal Infection; Neonatal SEPSIS
Keywords: Antibiotic switch therapy; Amoxicillin/clavulanic acid
MeSH Terms: conditions — Neonatal Sepsis | interventions — Amoxicillin-Potassium Clavulanate Combination; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized controlled non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral group (Active Comparator): After 48 hours of intravenous antibiotics eligible neonates will switch to amoxicillin/clavulanic acid suspension for the remaining 5 days. When the oral suspension is well tolerated neonates can be discharged from hospital.
  In order to investigate the pharmacokinetic profile of oral amoxicillin/clavulanic acid serum levels will be measured.
  Interventions: Drug: Amoxicillin Clavulanate
- Intravenous group (Active Comparator): Neonates will complete the full course of antibiotics of 7 days intravenously in hospital following local protocol.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — Dose 75 mg/kg/day, (3dd 25 mg/kg). Concentration amoxicillin/clavulanic acid: 4:1
  Arms: Oral group
Drug: Antibiotics — Intravenous antibiotic therapy following local protocol
  Arms: Intravenous group

SUMMARY:
Randomized controlled open-label non-inferiority trial comparing complete intravenous antibiotic treatment with a short iv. course followed by oral antibiotics in neonates (0-28 days) with probable bacterial infection.

Primary outcome:

- Bacterial re-infection within 28 days after finishing of antibacterial therapy.

Secondary outcome(s):

* Pharmacokinetic profile of oral amoxicillin/clavulanic acid
* Quality of life
* Cost-effectiveness
* Alterations in gut microbiome
* Use of molecular techniques for better detection of bacterial pathogens

DETAILED DESCRIPTION:
Neonates have a high antibiotic consumption because of their susceptibility for bacterial infections. Since the early diagnosis of bacterial infection in neonates is difficult, intravenous broad-spectrum antimicrobial therapy is usually started promptly after subtle symptoms. The majority of neonates become asymptomatic shortly after initiation; when infection is probable or proven by elevated inflammatory markers and/or a positive blood culture, intravenous antibiotics are administered for at least 7 days.

However, for neonates blood culture has a limited sensitivity. Therefore, the majority of neonates with probable infection are treated for a prolonged time with intravenous broad-spectrum antimicrobial therapy. In older children, intravenous antibiotics are often changed to oral antibiotics after cessation of symptoms and decreasing inflammatory parameters. This is not yet widely practised in neonates because of uncertainties in pharmacokinetics. Two explorative small studies from France and Italy into neonatal antibiotic switch therapy suggest that follow-up treatment with an oral antibiotic is promising; but the non-inferiority and safety was not yet properly addressed. Neonatal switch therapy, if proven to be safe and efficacious, would have a major impact on neonatal well-being, mother-to-child bonding and moreover costs.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (≥ 35+0 weeks, 0-28 days old, ≥ 2 kg)
* Probable bacterial infection defined as clinical symptoms and/or maternal risk factors and elevated inflammatory markers for which empiric broad-spectrum antibiotic treatment was initiated and needs to be continued for > 48 hours
* Clinically well
* Toleration of oral feeding without overt vomiting
* Signed informed consent

Exclusion Criteria:

* Proven bloodstream infection
* Absence of blood culture
* Severe localized infection (meningitis, osteomyelitis, necrotizing enterocolitis)
* Severe clinical sepsis (compromised circulation, need for mechanical ventilation)
* Continuous need for a central venous line
* Severe hyperbilirubinemia exceeding the exchange level
* Parents inability to administer medication
* Major congenital or syndromic anomalies

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 510 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Bacterial re-infection within 28 days after cessation of antibiotic treatment (within 35 days after initial presentation) | 0-35 days

SECONDARY OUTCOMES:
Duration of hospitalization | 0-35 days after birth
Percentage of re-admission | 0-35 days after birth
Total costs and cost-effectiveness | 0-35 days after birth
  Cost-effectiveness of intravenous to oral switch compared to a full course of antibiotics + possible extra costs due to early antibiotic switch
Difference in Quality of Life between oral and intravenous antibiotic treatment | 0-35 days after birth
  Two questionnaires on day 7 and 21 after admission, filled in by both parents. Data will be provided in a descriptive manner as no validated QoL questionnaires exist for neonates.
Time above MIC (T>MIC) of oral amoxicillin. | 0-7 days
  2 blood samples after administration of antibiotic suspension at different time points will be taken.
  Time above MIC (T>MIC) will be defined. Target MIC is 8 mg/liter.
Time above MIC (T>MIC) of oral clavulanic acid. | 0-7 days
  2 blood samples after administration of antibiotic suspension at different time points will be taken.
  Time above MIC (T>MIC) will be defined. Target MIC is 8 mg/liter.

CONTACTS AND LOCATIONS:
Overall Officials: Gerdien Tramper, Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (18):
- Netherlands (18):
  - Meander Medical Center, Amersfoort
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC-Sophia Children's Hospital, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Franciscus Vlietland, Schiedam
  - Haaglanden Medical Center, The Hague
  - Juliana Kinderziekenhuis-Haga Hospital, The Hague
  - Maxima Medisch Centrum, Veldhoven
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request through a repository and shared after consent of the principal investigator.

REFERENCES:
- [Derived] Keij FM, Kornelisse RF, Hartwig NG, van der Sluijs-Bens J, van Beek RHT, van Driel A, van Rooij LGM, van Dalen-Vink I, Driessen GJA, Kenter S, von Lindern JS, Eijkemans M, Stam-Stigter GM, Qi H, van den Berg MM, Baartmans MGA, van der Meer-Kappelle LH, Meijssen CB, Norbruis OF, Heidema J, van Rossem MC, den Butter PCP, Allegaert K, Reiss IKM, Tramper-Stranders GA. Efficacy and safety of switching from intravenous to oral antibiotics (amoxicillin-clavulanic acid) versus a full course of intravenous antibiotics in neonates with probable bacterial infection (RAIN): a multicentre, randomised, open-label, non-inferiority trial. Lancet Child Adolesc Health. 2022 Nov;6(11):799-809. doi: 10.1016/S2352-4642(22)00245-0. Epub 2022 Sep 9. PMID 36088952
- [Derived] Keij FM, Kornelisse RF, Hartwig NG, Mauff K, Poley MJ, Allegaert K, Reiss IKM, Tramper-Stranders GA. RAIN study: a protocol for a randomised controlled trial evaluating efficacy, safety and cost-effectiveness of intravenous-to-oral antibiotic switch therapy in neonates with a probable bacterial infection. BMJ Open. 2019 Jul 9;9(7):e026688. doi: 10.1136/bmjopen-2018-026688. PMID 31289068